CLINICAL TRIAL: NCT00659100
Title: A 3-Month, Open-Label, Pharmacy-Based, Actual-Use Trial in a Simulated Over-The-Counter (OTC) Environment to Assess Self-Selection and Consumer Use Patterns of Gabapentin 250 mg for Occasional Sleeplessness
Brief Title: A Trial to Assess Consumer Self-Selection and Use of Gabapentin for Occasional Sleeplessness in an Over-the-Counter Environment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A9451159
Record Dates: First submitted 2008-04-01; First posted 2008-04-16 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2011-04

CONDITIONS: Transient Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Gabapentin — Gabapentin 50 mg oral capsule 30 minutes before bedtime

SUMMARY:
The purpose of this study is to assess consumers' behaviors related to gabapentin self- selection and use, relative to warnings and directions for use, as described in the proposed over-the-counter (OTC) product label.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older with symptoms of sleeplessness
* Provided informed consent

Exclusion Criteria:

* Contraindications to use of gabapentin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1254 (Actual)
Dates: Start 2006-08; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who selected or purchased gabapentin for use (patients had symptoms consistent with indication and no contraindications) | Throughout Day 90
Subject compliance with directions for use (number of capsules per dose and the number of doses per day) | Throughout Day 90

SECONDARY OUTCOMES:
Adverse events | Duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (32):
- United States (32):
  - Pfizer Investigational Site, Anaheim, California
  - Pfizer Investigational Site, Bonita, California
  - Pfizer Investigational Site, Fallbrook, California
  - Pfizer Investigational Site, Hacienda Heights, California
  - Pfizer Investigational Site, La Mesa, California
  - Pfizer Investigational Site, Oceanside, California
  - Pfizer Investigational Site, Orange, California
  - Pfizer Investigational Site, San Dimas, California
  - Pfizer Investigational Site, Pembroke Pines, Florida
  - Pfizer Investigational Site, Weston, Florida
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Elk River, Minnesota
  - Pfizer Investigational Site, Northfield, Minnesota
  - Pfizer Investigational Site, Red Wing, Minnesota
  - Pfizer Investigational Site, Saint Louis Park, Minnesota
  - Pfizer Investigational Site, Holly Springs, Mississippi
  - Pfizer Investigational Site, Belton, Missouri
  - Pfizer Investigational Site, Independence, Missouri
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, Taos, New Mexico
  - Pfizer Investigational Site, Cary, North Carolina
  - Pfizer Investigational Site, Chapel Hill, North Carolina
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Pearland, Texas
  - Pfizer Investigational Site, Bountiful, Utah
  - Pfizer Investigational Site, Ogden, Utah
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Syracuse, Utah
  - Pfizer Investigational Site, West Valley City, Utah
  - Pfizer Investigational Site, Falls Church, Virginia
  - Pfizer Investigational Site, Richmond, Virginia

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9451159&StudyName=A%20Trial%20to%20Assess%20Consumer%20Self-Selection%20and%20Use%20of%20Gabapentin%20for%20Occasional%20Sleeplessness%20in%20an%20Over-the-Counter%20Environment